CLINICAL TRIAL: NCT01388101
Title: Real-time Diagnosis of Serum LECT 2 in Patient With Liver Cancer Using Electronic Antibody Sensor (e- Ab Sensor)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201007073R
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Liver Cancer
Keywords: LECT2
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LECT2 detection (Experimental): single-arm study: Electrosensing antibody probing system(e-AB sensor)
  Interventions: Device: Electrosensing antibody probing system (e- Ab sensor)

INTERVENTIONS:
Device: Electrosensing antibody probing system (e- Ab sensor) — Electrosensing antibody probing system (e- Ab sensor), which was developed for the rapid and sensitive detection of hapten, proteins, or viral antigen in medical samples, will be used for analyzing the interaction kinetics between specific anti- LECT2 and its antigen (LECT2 with liver cancer) present in the specimens of patients with liver cancer. The system incorporates the use of engineered semiconductive antibodies or virus in vertical and lateral chip (eAbchip) or lateral flow through (eAbsignal) formats. In electrosensing antibody probing, semiconductive antibodies are bound as a suitable electrosensing probe, which specifically and selectively binds targeted molecules (i.e. specific LECT2) in the test specimens.

SUMMARY:
To develop a real-time diagnostic technique with e- Ab sensor for specific LECT2 detection in clinical specimens of Hepatocellular carcinoma (HCC) patients, the investigators conduct a prospective clinical study. In comparison with results from direct sequencing of LECT2, the investigators evaluate the performance of e- Ab sensor, including reproducibility, sensitivity, specificity, and cross-reaction. With such technique, the investigators can obtain LECT2 information of HCC patients in cost-saving and time-saving way and can offer more individualized treatment for our patients.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most common types of cancer in the world. High cancer recurrence is still the major cause of death of HCC patients. The major poor prognostic factors included vascular invasion, high α-FP, large tumor size, or tumor satellitosis, etc. Among the various literature reports with multivariate analysis, vascular invasion of the tumor is the major contribution of high recurrence and poor survival. Therefore, identifying differentially expressed genes between vascular-invasion and non-vascular invasion of HCCs is important.

After suppression subtractive hybridization and microarray experiments, the investigators identified 20 differentially-expressed genes between vascular-invasive, and non-vascular invasive HCCs. One of the most interesting gene is leukocyte cell-derived chemotaxin 2 (LECT2). Further evaluation of the role of LECT2 on HCCs, the investigators found (1) Higher invasiveness, the lower of LECT2 gene expression in the HCC cell lines. (2) Conditioned medium with high LECT2 content will inhibit HCC invasion. (3) The invasion ability decreased in LECT2-overexpression hepatoma cell line. (4) In transendothelial cell migration assay, the investigators could observed invasion ability increased when LECT2 was knockdown in HCC cell line. (5) The lower expression of LECT2 gene in human HCCs correlate with higher tumor stage, early recurrence, and poor prognosis. (6) In vivo experiments revealed LECT2 can inhibit the ability of intravasation or metastatic ability of HCC.

Electrosensing antibody probing system (e- Ab sensor), which was developed for the rapid and sensitive detection of hapten, proteins, or viral antigen in medical samples, will be used for analyzing the interaction kinetics between specific anti- LECT2 and its antigen (LECT2 with liver cancer) present in the specimens of patients with liver cancer. The system incorporates the use of engineered semiconductive antibodies or virus in vertical and lateral chip (eAbchip) or lateral flow through (eAbsignal) formats. In electrosensing antibody probing, semiconductive antibodies are bound as a suitable electrosensing probe, which specifically and selectively binds targeted molecules (i.e. specific LECT2) in the test specimens. From assessment of the electric signature of semiconductive mutation-specific anti-LECT2 antibodies, the eABprobe could offer sensitive detection and precise quantification of specific LECT2.

To develop a real-time diagnostic technique with e- Ab sensor for specific LECT2 detection in clinical specimens of HCC patients, the investigators conduct a prospective clinical study. The investigators evaluate the performance of e- Ab sensor, including reproducibility, sensitivity, specificity, and cross-reaction. With such technique, the investigators can obtain LECT2 information of HCC patients in cost-saving and time-saving way and can offer more individualized treatment for our patients.

ELIGIBILITY:
Inclusion Criteria:

* The patients with liver cancer.
* The patients without liver cancer.

Exclusion Criteria:

1. Inmates, aboriginal peoples, pregnant women, mental patients, students, subordinates and other vulnerable groups.
2. Patients with malignant tumors.
3. Patients will be excluded if they couldn't sign the consent.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
The performance of e- Ab sensor | 1 Day
  In comparison with results from direct concentration of LECT2, we evaluate the performance of e- Ab sensor, including reproducibility, sensitivity, specificity, and cross-reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Chih Ho, MD,PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan